CLINICAL TRIAL: NCT01340287
Title: Effects of the Consumption of a Plant Sterols-enriched Dairy Fermented Product on Hypercholesterolemia Management in Hypercholesterolemic Adults
Brief Title: Effect of the Consumption of a Fermented Milk Enriched With Plant Sterols
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU281
Record Dates: First submitted 2011-04-21; First posted 2011-04-22 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Hypercholesterolemia
Keywords: Plant sterol; Hypercholesterolemia; diet; dairy; isoprostanes; Midly hypercholesterolemic subjects
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 = Tested product (Active Comparator)
  Interventions: Dietary Supplement: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols).
- 2 = Control product (Sham Comparator)
  Interventions: Dietary Supplement: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters

INTERVENTIONS:
Dietary Supplement: 1- plain low-fat dairy fermented product (drinkable) enriched with plant sterols-esters (1,6g /day equivalent as free sterols). — 1 = Intervention 1 (1 test product/day)
  Arms: 1 = Tested product
Dietary Supplement: 2- plain low-fat dairy fermented product (drinkable) without plant sterols-esters — 2 = Intervention 2 (1 control product/day)
  Arms: 2 = Control product

SUMMARY:
The purpose of this study is to investigate the cholesterol lowering effect of a drinkable low fat fermented milk enriched with plant sterol after 3 and 6 weeks of daily consumption in midly hypercholesterolemic people not treated by statins.

ELIGIBILITY:
Inclusion Criteria:

* male/female subject,
* aged from 21 to 75 years,
* BMI between 19 and 30 kg/m2,
* LDL-cholesterol plasma level between 130 and 190 mg/dL without statin monotherapy,
* stabilized hypercholesterolemia,
* accepting to follow the dietary recommendations advisable for hypercholesterolemic patient (NCEP-ATP III guidelines),
* used to consume dairy products,
* effective contraceptive methods used for female subjects,
* having given written consent to take part in the study

Exclusion Criteria:

* subject with plasma triglycerides (TG) levels ≥ 350 mg/dL,
* having experienced any cardiovascular event in the last 6 months,
* taking any hypocholesterolemic treatment,
* diabetic subject (type I and type II),
* smoking strictly more than 10 cigarettes / day,
* heavy alcohol intake (> 40 g / day for men ; > 30 g / day for women),
* presenting known allergy or hypersensitivity to milk proteins,
* known soy allergy,
* refusing to stop the consumption of plant sterols-enriched products (other than the studied product),
* receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters,
* receiving a transplant and under immunosuppressor treatment,
* currently involved in a clinical trial or in an exclusion period following participation in another clinical trial,
* in a situation which in the investigator's opinion could interfere with optimal participation in the present study or could constitute a special risk for the subject,
* with any kind of disease likely to interfere with the evaluation of efficiency or safety of the product,
* for female subject: pregnancy, breast feeding or intention to be pregnant during the study or subject likely to change her contraceptive method during the study

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 168 (Actual)
Dates: Start 2008-07; Primary Completion 2009-05 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Renstar Medical Research, Ocala, Florida, United States